CLINICAL TRIAL: NCT03298789
Title: Acute Effects of Static Stretching in Warm-up on Muscular Performance of Football Players
Brief Title: Acute Effects of Static Stretching in Warm-up
Acronym: AESSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Primorska (Other)
Collaborators: S2P, Science to Practice, Ltd. (Other); Motus Melior, Ltd. (Unknown)
Responsible Party: Principal Investigator, Nejc Sarabon, Assoc. Prof. Dr. Sc., University of Primorska
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UP-FVZ-StretchingEffects
Record Dates: First submitted 2017-08-03; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Only Healthy Participants Are Included in the Study
Keywords: static stretching; muscle power; countermovement jump; dynamometry; warm up; force plate

STUDY DESIGN:
Intervention Model Description: 19 subjects will be devided into two groups. The first group will conduct the control condition on Saturday and the second group will conduct the experimental condition on Sunday. One week later, the subjects will undergo the second visit, each group of subjects performing the opposite condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental condition (Experimental): 7 series of static stretching will be conducted in the experimental condition. Activation exercises will be performed after 7th series of static stretching.
  Interventions: Other: Activation exercise; Other: 7 series of static stretching
- Control (Other): 7 series of static stretching will be conducted in the control condition.
  Interventions: Other: 7 series of static stretching

INTERVENTIONS:
Other: Activation exercise — Two series of 4 activation exercise will be included in the intervention.
  Arms: Experimental condition
Other: 7 series of static stretching — 7 series of 4 20 seconds static stretches will be conducted.

SUMMARY:
In this study the investigators want to address acute effects of warm-up and static stretching on short-term muscular performance of football players. Static stretching exercises are often used in the first part of a training session or before a football match in order to increase sports performance and to decrease risk of injuries. Since there is a lot of scientific evidence that demonstrates static stretching can improve short-term muscle performance, the aim of researchers is to discover the size and the duration of negative effects and, additionally, whether these effects can be eliminated with activation exercises. Nineteen 14 years old football players will be included in a cross-over study design.

In the control condition the participants will perform 5 minutes of aerobic warm-up (stepping on the stair) and then 7 series of 20-seconds static stretching of quadriceps femoris, hamstrings, hip adductors and triceps surae.

Maximal power and jump height of the countermovement jump will be tested in between every series. Thus, parameters of countermovement jump will be monitored at the beginning, after warm-up, after each series of static stretching, 7.5 minutes after 7th static stretching series and 15 minutes after 7th static stretching series.

Parameters of dynamometry (relative maximal torque [Nm/kgBM] and rate of torque developement [Nm/s/kgBM] will be monitored at the beginning, after warm up, 7.5 minutes after last series of static stretching and 15 minutes after last series of static stretching.

Maximal range of motion will be monitored at the beginning, after warm up, during every series of static stretching, after last series of static stretching, 7.5 minutes after last series of static stretching and 15 minutes after last series of static stretching.

In the second condition (experimental) all the tasks are the same, the only difference is that the subjects must perform post-activation potentiation exercises after last series of static stretching.

We hypothesize that muscular performance will be impaired to a statistically significant level after 7th series of static stretching. Second hypothesis is that negative effects will not last longer than 15 minutes and the last hypothesis is that static stretching induced negative effects can be nullified with activation exercises.

DETAILED DESCRIPTION:
Stretching exercises are often used in warm-up to increase footballer's performance and to decrease risk of injury. The main aim of these exercises is to increase maximal active range of motion. Different types of stretching exercises are being used: ballistic, dynamic, static, eccentric flexibility training and proprioceptive neuromuscular facilitation. All of them are usually used in football training sessions in order to increase short-term range of motion and to decrease associated risk of injuries. Simic, Sarabon and Markovic (2013) in their meta-analysis reported that static stretching can have negative acute effects, which is not in line with general thinking, that static stretching in warm-up can have positive effects on sports performance.

Post-activation potentiation is a phenomenon, which is induced by loading the muscle to increase the recruitment of motor units. Since static stretching can have negative effects on muscle performance (maximal strength, power) the researchers hypothesize, that the effects can be eliminated with this type of activation exercises.

In this study the researchers want to measure acute effects of warm-up and static stretching on maximal range of motion, maximal torque and maximal rate of torque of adductors (dynamometer) and maximal power and height of countermovement jump (force plate) of football players. Since there is many scientific evidence that shows that static stretching can improve short-term muscle performance, our aim is to discover the size and the duration of negative effects and if they can be eliminated with post-activation potentiation exercises. In the cross-over study design 19 football players of age 14 will be included.

In the first condition (control) the participants will perform 5 minutes of aerobic warm-up (stepping on the stair) and then 7 series of 20-seconds bilateral static stretching of hamstrings, adductors and triceps surae (with knee extended). Quadriceps femoris will be stretched unilaterally, each muscle 20 seconds. Summary of all stretches in one series is 80 seconds. Maximal range of motion of hip abduction and hip flexion (seat and reach test) and dorsal flexion will be measured at the beginning, after warm up, during each series of static stretching, after last series of static stretching, 7.5 minutes after last series of static stretching and 15 minutes after last series of static stretching.

Maximal power [W/kg] and height [m] of the countermovement jump will be monitored with force plate at the beginning, after warm up, after each series of static stretching, 7.5 minutes after last series of static stretching and 15 minutes after last series of static stretching.

On dynamometer will be conducted 2 maximal explosive voluntary contractions of adductors muscles. Relative maximal torque [Nm/kgBM] and rate of torque developement [Nm/s/kgBM] will be measured at the beginning, after warm up, after last series of static stretching, 7.5 minutes after last series of static stretching and 15 minutes after last series of static stretching.

In the second condition (experimental) all the tasks are the same, the only difference is that the subjects must conduct activation exercises after last series of static stretching.

Activation exercises are consisted of 2 series of 4 exercises. The first series (slow series) starts with 8 lifts onto toes (dorsal flexion) with knees extended, than continues with 8 deep squats and 8 hip thrust and then terminates with four 4-seconds lasting maximal voluntary contraction of adductors with knees extended and with soft ball between the ankles. The second series (explosive) commences with 8 maximal vertical jumps conducted just with ankles, and then continues with 8 maximal countermovement jumps and 8 explosive hip thrusts. It finishes with 8 maximal explosive and 2 seconds lasting voluntary contractions of hip adductors with knees extended and with soft ball between the ankles.

The researchers hypothesize that muscular performance (maximal power and height of the countermovement jump, maximal torque and rate of torque developement of adductors muscles) will be impaired after 7 series of static stretching. Second hypothesis is that negative effects will not last longer than 15 minutes and the last hypothesis is that static stretching induced negative effects can be eliminated with sets of activation exercises.

Statistical analysis will be performed in SPSS (SPSS Statistics 22, IBM, New York). T-test, 1-way and 2-way repeated measures ANOVA will be used to confirm the differences between average values.

ELIGIBILITY:
Inclusion Criteria:

* football players, man

Exclusion Criteria:

* injuries, last 12 months

Ages: 12 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2017-07-23 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Muscle Performance | 1 week
  Maximal and explosive strength of adductors, maximal power during countermovement jump

SECONDARY OUTCOMES:
Maximal power during countermovement jump | 1 week
  Relative maximal power during countermovement jump on force plate (W/kg)
Jump Height | 1 week
  Maximal height of countermovement jump on force plate (m)
Relative maximal torque of adductors on dynamometer (Nm/kgBM) | 1 week
  Maximal voluntary contraction of adductors will be performed on dynamometer.
Rate of torque developement (Nm/s/kgBM) | 1 week
  Rate of torque developement were monitored during Explosive maximal voluntary contraction of adductors performed on dynamometer.
Maximal range of motion (cm) | 1 week
  Maximal range of passive motion (bilaterally performed: seat&reach, hip abduction, dorsal foot flexion - for all, knees extended)

CONTACTS AND LOCATIONS:
Overall Officials: Nejc Sarabon, PhD, Study Director — University of Primorska, Faculty of Health Studies, Izola, Slovenia
Locations (1):
- Faculty of Health Studies, University of Primorska, Izola, Polje 42, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided